CLINICAL TRIAL: NCT01599676
Title: "Effect of Citrulline Supplementation on Muscle Strength in Elderly Institutionalized Subjects Undergoing an Exercise Training Programme. "
Brief Title: Citrulline, Exercise Training and Muscle Strength in the Elderly
Acronym: CITREX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AOM 09008; N° IDRCB: 2010-A002346-33 (Other Grant/Funding Number: IDRCB: 2010-A002346-33)
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Elderly Patients
Keywords: Citrulline; protein-energy malnutrition; amino acids; muscle strength; resistance training
MeSH Terms: conditions — Protein-Energy Malnutrition | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Not essential amino acid (Sham Comparator): Non essential amino acid:
  The subjects will have a regimen of high-intensity progressive resistance training of the knee extensors 3 days per week for 12 weeks. The subjects will receive 1 unit of an equivalent quantity of nonessential amino acids (alanine, aspartate, glycine, serine, histidine and proline in equimolar quantity) isonitrogenous to 10 g of citrulline, once in the morning for 12 weeks.
  Interventions: Dietary Supplement: Non essential amino acid
- Citrulline (Experimental): The subjects will have a regimen of high-intensity progressive resistance training of the knee extensors 3 days per week for 12 weeks. The subjects will receive citrulline 10 g/day orally in the morning for 12 weeks.
  Interventions: Dietary Supplement: Citrulline

INTERVENTIONS:
Dietary Supplement: Citrulline — The subject will receive citrulline 10 g/day orally in the morning for 12 weeks.
  Other Names: Dietary supplement Citrulline
  Arms: Citrulline
Dietary Supplement: Non essential amino acid — Non essential amino acid supplementation
  Other Names: Non essential amino acid supplementation
  Arms: Not essential amino acid

SUMMARY:
The aim of this study is to assess the effect of citrulline supplementation on muscle strength in elderly institutionalized subjects undergoing a resistance exercise training program. The primary endpoint is the outcome of maximum strength of knee extensor muscles.

DETAILED DESCRIPTION:
Maintaining muscle strength is mandatory for elderly persons to keep autonomy. Resistance exercise increases muscle strength in old and very old subjects, but there seems to be little effect on muscle mass. Citrulline is an amino acid that stimulates muscle protein synthesis, but its effect on muscle strength and mass remains to be determined. The aim of this study is to assess the effect of citrulline supplementation on muscle strength in elderly institutionalized subjects undergoing a resistance exercise training program.

All the subjects (84) will undergo a resistance exercise training program for 12 weeks. The subjects will have a regimen of high-intensity progressive resistance training of the knee extensors 3 days per week. These muscle groups were chosen because of their importance in functional activities. The subjects will be randomized into two groups. An intervention group will receive orally citrulline at 10 g/day, and a control group will receive an isonitrogenous amount of nonessential amino acids (alanine, aspartate, glycine, serine, histidine and proline in equimolar quantity). During the 12 weeks of supplementation, clinical tolerance will be evaluated. Strength testing will be repeated every two weeks for 12 weeks. The primary endpoint is the outcome of maximum strength of knee extensor muscles. Fat-free mass (DEXA), gait velocity, timed get up and go, spontaneous physical activity (activity monitors), nutritional status (weight, albuminemia, TRANSTHYRETINEMIA) and quality of life will be measured at inclusion and at the end of the study. The number of falls during the study will be recorded.

ELIGIBILITY:
INCLUSION CRITERIA:

* Aged over 75 years
* Able to walk at least 6 meters without human assistance.

EXCLUSION CRITERIA:

* Moderate to severe cognitive disorders (MMSE < 20)
* Severe malnutrition (BMI < 18 or weight loss > 10 % in 1 month or > 15 % in 6 months, or albuminemia < 30 g/L),
* Inflammation (CRP > 30 mg/L),
* Severe renal failure (creatinine clearance < 30 mL/mn),
* Stage 4 cardiac failure,
* Respiratory failure,
* Corticoid treatment,
* Participation in another trial

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Maximum strength of knee extensor muscles | 12 weeks
  Strength testing will be repeated every two weeks for 12 weeks

SECONDARY OUTCOMES:
Fat-free mass | 12 weeks
  Fat-free mass was measured by DEXA

CONTACTS AND LOCATIONS:
Overall Officials: Christian Aussel, PHD, Study Director — Assistance Publique Hopitaux de Paris
Locations (1):
- HOPITAL BICHAT Claude Bernard, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided